CLINICAL TRIAL: NCT02334501
Title: An Open-Label, 2-Period, Fixed Sequence Study to Evaluate the Effect of Lansoprazole on the Pharmacokinetics of Neratinib in Healthy Subjects
Brief Title: Open-label PK Study to Evaluate Lansoprazole and Neratinib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PUMA-NER-0101
Record Dates: First submitted 2014-10-21; First posted 2015-01-08 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — Lansoprazole; neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment A (Period 1) and Treatment B (Period 2) (Experimental): Treatment A (240mg Neratinib x1) Treatment B (30mg Lansoprazole X 7 days + 240mg Neratinib x1)
  Interventions: Drug: Lansoprazole; Drug: Neratinib

INTERVENTIONS:
Drug: Lansoprazole
Drug: Neratinib

SUMMARY:
This is an open label, 2-period, fixed-sequence study in 15 healthy adult subjects under fed conditions. To evaluate the effect of multiple doses of lansoprazole on the absorption and pharmacokinetics (PK) of a single dose of neratinib in healthy subjects.

DETAILED DESCRIPTION:
This is an open label, 2-period, fixed-sequence study in 15 healthy adult subjects under fed conditions. On Day 1 of Period 1 (Treatment A), a single oral dose of neratinib will be administered followed by PK sampling for 72 hours. In Period 2 (Treatment B), multiple oral doses of lansoprazole will be administered once daily for 7 consecutive days with a single oral dose of neratinib administered on Day 5. PK sampling for neratinib will be taken for 72 hours following neratinib dosing on Day 5. The washout period will be at least 14 days between each neratinib dose.

ELIGIBILITY:
Inclusion Criteria:

Healthy, adult, men or women, 18 to 55 years of age, inclusive, at screening. Body Mass Index ≥ 18.5 and ≤ 32.0 kg/m2 at screening. Non to moderate smokers (up to 10 cigarettes a day for at least 3 months prior to screening).

Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or 12-lead electrocardiograms (ECGs), as deemed by the principal investigator (PI).

Women of childbearing potential: either be sexually inactive (abstinent) for 14 days prior to the first dose and for at least 28 days following the last dose or be using one of the protocol-specific birth control methods.

Exclusion Criteria:

Acute disease state (eg, nausea, vomiting, fever, or diarrhea) within 7 days prior to the first dose of study drug.

History or presence of alcoholism or drug abuse within the past 2 years prior to screening.

History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds (eg, proton-pump inhibitors [PPIs]).

Women who are pregnant or lactating. Positive results at screening for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus.

Unable to refrain from or anticipates the use of:

* Any drug, including prescription and nonprescription medications, herbal remedies, or vitamin supplements (including proton-pump inhibitors) beginning 14 days prior to the first dose of study drug and throughout the study. Acetaminophen (up to 2 g per 24 hour period) and/or loperamide (up to 6 mg per 24 hours) may be permitted during the study at the direction of the PI.
* Any drugs known to be significant inducers of cytochrome p450 enzymes and/or P glycoprotein, including St. John's Wort, for 28 days prior to the first dose of study drug and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of PK/pharmacodynamics interaction with study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) of neratinib with and without lansoprazole | 0, 0.5, 1, 2, 2.75, 3.5, 4.25, 5, 5.75, 6.5, 7.25, 8, 10, 12, 24, 32, 48, 60, and 72 hours post-dose
  The area under the plasma concentration-time curve, from time 0 to the last measurable nonzero concentration, as calculated by the linear trapezoidal method.
AUC(0-inf) of neratinib with and without lansoprazole | 0, 0.5, 1, 2, 2.75, 3.5, 4.25, 5, 5.75, 6.5, 7.25, 8, 10, 12, 24, 32, 48, 60, and 72 hours post-dose
  The area under the plasma concentration-time curve from time 0 extrapolated to infinity. AUC(0-inf) is calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Cmax of neratinib with and without lansoprazole | 0, 0.5, 1, 2, 2.75, 3.5, 4.25, 5, 5.75, 6.5, 7.25, 8, 10, 12, 24, 32, 48, 60, and 72 hours post-dose
  Maximum observed concentration.

SECONDARY OUTCOMES:
Number of participants with adverse events | over 4 week study period
  Safety endpoints will include all AEs, physical examinations, vital signs, 12-lead electrocardiograms (ECGs), and clinical laboratory tests (hematology, serum chemistry, and urinalysis).

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States